CLINICAL TRIAL: NCT03301896
Title: A Phase I/Ib, Open-label, Multi-center Dose-escalation and Dose-expansion Study of the Safety and Tolerability of Intra-tumorally Administered LHC165 Single Agent and in Combination With PDR001 in Patients With Advanced Malignancies
Brief Title: Study of the Safety and Efficacy of LHC165 Single Agent and in Combination With PDR001 in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLHC165X2101
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumors
Keywords: Phase I; LHC165; PDR001; intratumoral injection; abscopal; checkpoint inhibitor; programmed cell death; PD-1; TLR-7; toll-like receptor; melanoma; head and neck
MeSH Terms: conditions — Melanoma | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LHC165 single agent (Experimental): LHC165 intratumoral injection given alone
  Interventions: Drug: LHC165
- LHC165 in combination with PDR001 (Experimental): LHC165 intratumoral injection given with PDR001 infusion
  Interventions: Drug: LHC165; Biological: PDR001

INTERVENTIONS:
Drug: LHC165 — LHC165 intratumoral injection
Biological: PDR001 — PDR001 infusion
  Arms: LHC165 in combination with PDR001

SUMMARY:
The purpose of this trial was to explore the clinical utility of two investigational agents in patients with advanced cancer.

This was a multi-center, open-label Phase I/Ib study. The primary objectives of the trial were:

* To characterize the safety and tolerability of intratumoral LHC165 in patients with solid tumors as a single agent and in combination with PDR001
* To determine and evaluate the maximum tolerated dose (MTD)/recommended dose (RD) for LHC165 as a single agent and in combination with PDR001

DETAILED DESCRIPTION:
This was a multi-center, open-label Phase I/Ib study. The study consisted of four dose escalation parts and two dose expansion parts testing LHC165 as a single agent or LHC165 in combination with PDR001. The dose escalation parts estimated the Maximum Tolerated Dose (MTD) and/or Recommended Dose for Expansion (RDE) and were planned to test two different dosing schedules for LHC165 single agent (Group A and B) and LHC165 in combination with PDR001 (Group C and D).

The dose expansion parts of the study were planned to use the MTD/RDE for each the LHC165 single agent (Group E) and LHC165 in combination with PDR001 (Group F), determined in the respective dose escalation parts to assess the activity, safety and tolerability of LHC165 as a single agent or LHC165 in combination with PDR001 in patients with specific types of solid tumors.

The study was terminated due to business reasons. Groups B, D and E were not opened for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any procedures unless considered standard of care.
* Adult men and women (≥ 18 years of age) with histologically confirmed diagnosis of metastatic and/or advanced solid tumors not amenable to curative treatment by surgery.
* Patients must be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Dose escalation: Patients with accessible tumors and with measurable disease as determined by RECIST 1.1 and have progressed despite standard treatment or are intolerant of standard treatment, or for whom no standard treatment exists.
* Dose expansion: Patients with advanced/metastatic solid tumors: HNSCC, melanoma, accessible tumors and visceral tumors (LHC165 combination with PDR001 only). Patients must have measurable disease as determined by RECIST 1.1 and have progressed despite standard treatment or are intolerant to standard treatment, or for whom no standard treatment exists• Patients must have at least two sites of disease amenable to biopsy.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion Criteria:

* Presence of symptomatic or uncontrolled central nervous system (CNS) metastases requiring local CNS-directed treatment.
* Patients diagnosed with hematological malignancies.
* Patients with prior stem cell transplants.
* Patients previously treated with TLR-7/8 agonist treatment.
* History of primary immunodeficiency
* Patients who discontinued prior anti-PD-1/PD-L1 therapy due to an anti-PD-1/PD-L1-related toxicity.
* Malignant disease, other than that being treated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Escalation: Incidence of Dose-limiting Toxicities (DLTs) in Cycle 1 | day 28
  Dose Limiting Toxicity Evaluation Period
Escalation and Expansion: Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs), including changes in laboratory parameters, vital signs, electrocardiograms (ECGs) | 24 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 and iRECIST | 24 months
Best Overall Response (BOR) per RECIST 1.1 and iRECIST | 24 months
Progression-Free Survival (PFS) per RECIST 1.1 and iRECIST | 24 months
Duration of Response (DOR) per RECIST 1.1 and iRECIST | 24 months
Disease Control Rate (DCR) per RECIST 1.1 and iRECIST | 24 months
Serum concentration profiles of LHC165 as a single agent: Cmax | 24 months
Serum concentration profiles of LHC165 in combination with PDR001 and derived PK parameters: Cmax | 24 months
Serum concentration profiles of PDR001 in combination with LHC165 and derived PK parameters: Cmax | 24 months
Serum concentration profiles of LHC165 as a single agent: AUC | 24 months
Serum concentration profiles of LHC165 in combination with PDR001 and derived PK parameters: AUC | 24 months
Serum concentration profiles of PDR001 in combination with LHC165 and derived PK parameters: AUC | 24 months
Serum concentration profiles of LHC165 as a single agent: Tmax | 24 months
Serum concentration profiles of LHC165 in combination with PDR001 and derived PK parameters: Tmax | 24 months
Serum concentration profiles of PDR001 in combination with LHC165 and derived PK parameters: Tmax | 24 months
Presence and titer of anti-PDR001 antibodies | 24 months
Change from baseline in tumor infiltrating lymphocytes in injected and distal tumor specimens | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Parikh, MD, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (2):
  - UCLA, Los Angeles, California
  - MD Anderson Cancer Center, Houston, Texas
- Novartis Investigative Site, Wilrijk, Belgium
- Novartis Investigative Site, Ulm, Germany
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18030
- See also: Plain Language Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1546